CLINICAL TRIAL: NCT07335809
Title: Study on the Impact of Nursing Interventions Based on the ABC-X Model on Psychological Resilience and Family Functioning in Patients After Total Knee Arthroplasty
Brief Title: Impact of ABC-X Model Nursing on Psychological Resilience and Family Function in TKA Patients
Status: Not yet recruiting | Type: Observational
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2025-219
Record Dates: First submitted 2025-12-15; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Implement nursing interventions based on the ABC-X model — Establish a Nursing Team Based on the ABC-X Model
  Implement the Nursing Intervention Plan:
  1. A - Stressor Assessment, including physiological assessment, assessment of life challenges, and evaluation of the social support network.
  2. B - Coping Resources, involving organizing medical system resources, individual internal resources, and family and social resources.
  3. C - Cognitive Appraisal: Use open-ended questioning to help patients understand the normality of stress responses, reduce fear of negative emotions, and minimize self-blame.
  4. X - Crisis Outcome, assessing the patient's emotional state, behavioral responses, physiological reactions, and family functioning.
  The intervention will be conducted over a period of 6 months.

SUMMARY:
The ABC-X model is a systematic intervention approach based on stress source analysis and adaptation theory. It emphasizes the dynamic interaction between stressors (A), coping resources (B), cognitive appraisal (C), and crisis outcomes (X). By systematically assessing patients' psychosocial stress, integrating family and social support resources, and optimizing disease cognition, it helps patients and their families alleviate psychological pressure and cope with disease challenges. This study aims to explore the impact of nursing interventions based on the ABC-X model on coping styles and family functioning in patients after total knee arthroplasty.

DETAILED DESCRIPTION:
Total Knee Arthroplasty (TKA) is primarily indicated for patients with knee joint diseases that are unresponsive to conservative treatment and significantly impair daily life and work, such as osteoarthritis, rheumatoid arthritis, traumatic arthritis, osteonecrosis, or other inflammatory joint conditions. It is one of the widely used and well-established surgical procedures in the field of orthopedics. This surgery can effectively alleviate pain, correct joint deformities, and restore joint function. However, TKA may still be associated with various postoperative complications. Coupled with the prolonged off-hospital rehabilitation period, patients often exhibit insufficient compliance and limited coping strategies, which can adversely affect their postoperative recovery outcomes. Current routine nursing care primarily focuses on consolidating surgical outcomes, preventing complications, and promoting functional recovery. While it helps improve patients' daily activity levels and facilitates postoperative rehabilitation, it lacks systematic intervention in addressing patients' psychological stress, family support, and the integration of social resources. Moreover, patients often experience varying degrees of impaired self-care ability in the short term after surgery, necessitating reliance on family members for daily assistance. Therefore, when patients transition from hospital to family and social life, providing them with a professional and multifaceted nursing model is crucial, as it directly influences the speed and quality of their recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for knee osteoarthritis as outlined in the Guidelines for Diagnosis and Treatment of Osteoarthritis (2018 Edition)[6], with confirmation by imaging examination;
2. Age 30-65 years;
3. Meet the surgical indications of our hospital and be a first-time candidate for unilateral TKA;
4. Normal neurological and cognitive function, with stable vital signs;
5. Family members have signed the informed consent form.

Exclusion Criteria:

1. Presence of lower limb movement impairments;
2. Accompanied by severe complications;
3. Infectious diseases or severe immune system disorders;
4. Other acute and critical illnesses;
5. History or presence of mental dysfunction;
6. Language or communication disorders.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 117 patients who underwent TKA for knee osteoarthritis from July 2025 to July 2026 were selected as the study subjects.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative recovery effectiveness | The intervention will be conducted over a period of 6 months.
  Postoperative recovery effectiveness: Six months after surgery, the modified Macnab criteria are used for therapeutic evaluation: Excellent indicates complete symptom relief with return to normal daily life and work; Good indicates mild symptoms with slight limitations on daily activities, without adverse effects on daily life and work; Fair indicates significant symptom relief but with limitations on daily activities and adverse effects on daily life and work; Poor indicates no improvement or worsening of symptoms before and after treatment.
Psychological resilience | Intervention will take place within 6 months.
  Psychological resilience：Evaluated using the Resilience Scale (CD-RISC), which has a Cronbach's α coefficient of 0.875, including three dimensions: strength (10 items, 40 points), optimism (8 items, 32 points), and 韧性 (7 items, 28 points). Each item is scored from 0 to 4 points, with a total score of 100 points, with higher scores indicating better psychological resilience.
Self-care ability | Intervention will take place within 6 months
  The Self-Care Ability Scale (ESCA) was used for evaluation, with a Cronbach's α coefficient of 0.86~0.92. It consists of 4 dimensions and 43 items, with each item scored on a scale of 0 to 4 points. The total score ranges from 0 to 172, with higher scores indicating stronger self-care ability.
Rehabilitation exercise adherence | Intervention will take place within 6 months
  The Functional Exercise Adherence Scale for Orthopedic Patients was used for assessment. This scale consists of 3 dimensions and 15 items, covering exercise adherence related to physical aspects, psychological aspects, and active learning. A 1-5 point Likert 5-point rating scale is used, with a total score of 75 points. Scores <20 points, 20-55 points, and ≥55 points respectively indicate low adherence, partial adherence, and high adherence.
Family functions | Intervention will take place within 6 months
  The Family Function Assessment Scale (APGAR) was used for evaluation, with a Cronbach's α coefficient of 0.856. It consists of 5 items: cooperativeness, adaptability, emotional quality, maturity, and intimacy. Each item is scored out of 10, with higher scores indicating better family function.

IPD SHARING:
Plan to Share IPD: Undecided